CLINICAL TRIAL: NCT03100682
Title: Prevention of Human Papillomavirus (HPV) Infection in Paediatric Kidney and Liver Transplant Recipients and in Paediatric Patients With Advanced Chronic Kidney Disease: a Prospective, Observational Multi-centre Vaccine Surveillance Study (HPVaxResponse Study)
Brief Title: Prevention of Human Papillomavirus (HPV) Infection in Paediatric Kidney and Liver Transplant Recipients and in Paediatric Patients With Advanced Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, PD Dr. med. Britta Hoecker, Privatdozentin Dr. med. Britta Hoecker, University Hospital Heidelberg
Other Study IDs: HPVaxResponse Study
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Paediatric Kidney or Liver Transplantation; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum rest material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to their immunosuppressive therapy, solid-organ transplant (SOT) recipients bear a 10 to 100 times higher risk of human papillomavirus (HPV)-associated malignancies than healthy individuals. The objectives of this observational, non-interventional multi-national, multi-centre research project are to gain an insight into current HPV vaccination strategies and to investigate the immune response to different routinely administered HPV vaccines in European paediatric SOT candidates and immunocompromised transplant recipients, enabling patients at risk of vaccination failure to be identified.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric Kidney and/or Liver transplant recipients
* Paediatric patients with CKD
* Who receive HPV vaccination according to country-specific vaccine schedule

Exclusion Criteria:

* No HPV vaccination according to country-specific vaccine schedule
* No written informed consent

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric Kidney and/or Liver transplant recipients Paediatric patients with CKD
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-03-18 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Immune Response to HPV vaccine | Change of immune response from baseline (prior to vaccination) to 4-12 weeks after vaccination and to 18+- 3 months after vaccination will be assessed.
  HPV vaccine antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Britta Hoecker, MD, Principal Investigator — University Children's Hospital of Heidelberg
Locations (1):
- University Children's Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided